## **CONFIDENTIAL**

# Case Report Form

Clinical Trial Protocol No. URSO – 003

Version 2, dated 17 August 2022

Multi-Center, randomized, control, phase IV trial to compare the efficacy & safety of Ursoplus® capsules (UDCA 250mg & Silymarin 140mg) versus UDCA alone versus Placebo among Compensated Chronic Liver Diseased Patients

| Please use a ball point Blue pen | |
|----------------------------------|------------------------|
| Investigator's Name and Address: | |
| Center N°: | |
| Patient's N°: | Patient's<br>Initials: |

**Property of Minapharm Pharmaceuticals** 

May not be used, divulged, published or otherwise disclosed Without the prior consent of Minapharm Pharmaceuticals

| Patient's<br>Nº: | | Patient's<br>Initials: | |
|---|---|---|---|
| General instructions: | | | |
| | <ol> <li>A CRF must be completed for each study participant who is successfully<br/>enrolled (successfully screened)</li> </ol> | | |
| 2- Please v<br>FORM | <ul> <li>Please write legibly upper case/capital letter is preferred e.g. CASE REPORT<br/>FORM</li> </ul> | | |
| 3 All entr | 3 All entries must be made preferably in blue ballpoint pen | | |
| 4- Do not | 4- Do not leave any question unanswered. | | |
| If the a | nswer to a question is unl | known/ for missing information | on. |
| Please | Please enter: NA - if data is not applicable or not available. | | |
| | | NK - if information is | s unknown. |
| | | ND - if procedure no | ot done |
| re- ente<br>correction<br>event or<br>Re-ente | r the data immediately abon. However, If you make medication / non – drug r the data in the space be | ke through original entry (e. gove the old entry, and initial e an error on the description therapy, please strike throughow the start date, and initial ite – out or obliterate informatics. | and date the for adverse gh original entry. I and date the |
| reports of must be | or clinic /hospital records | atient number and initials in are attached to the CRF, the with a black marker and the | e patient name |
| 7- Use lea | iding "0's" to complete en | tire field. | |
| 8- All CRF in the st | . • | d and signed by the investiga | ator participating |
| 9- All text a | and explanatory commen | ts should be brief | |
| 10-Answer | every question explicitly; | do not use ditto marks | |
| and accurate | data. I confirm that the st<br>any protocol amendments | plied in this case record forn<br>udy was conducted in accord<br>and that written informed co | dance with the |

Investigator's Signature:

Date of signature:

| Patient's | Patient's | Screening Visit |
|-----------|-----------|------------------|
| Nº: | Initials: | Initiation Visit |

#### **Numeric fields**

- 1- Enter only 1 digit in each box, with a leading 0 when necessary
- 2- Record all values in the unites indicated on the CRF

## Confidentiality

Patients must only be identified by the subject identification ID (Center number, Patient number

## **Adverse Event Log/Concomitant Medication Log**

If additional pages of adverse event and / or concomitant medication log are required, please make a photocopy of a blank adverse Event log / concomitant medication log and complete the information. The original page will be sent to data management and a photocopy retained at Minapharm and investigator site

#### **Dates**

- 1- All dates are to be reported in the format DD/MMM/YYYY
- 2- The month is to be reported as the first three characters of the month, e.g. 01/AUG/2012 the month abbreviations are as follows:

| January | = | Jan | May | = | May | September | = | Sep |
|----------|---|-----|--------|---|-----|-----------|---|-----|
| February | = | Feb | June | = | Jun | October | = | Oct |
| March | = | Mar | July | = | Jul | November | = | Nov |
| April | = | Apr | August | = | Aug | December | = | Dec |

3- In the absence of a precise date for an event or therapy that precedes the participant's inclusion into the study, a partial date may be recorded by recording "NK" in the fields that are unknown e.g. where the day and month are not clear, the following may be entered into the CRF:

| 0 | 0 | М | Α | R | 2 | 0 | 0 | 9 |
|---|---|---|-----|---|---|----|----|---|
| D | D | Ν | 1MI | M | | YY | ΥY | |

## **Center Numbering:**

Enter the center number (2 digits),

- Research Center of Air Force Specialized Hospital = 01
- ➤ Helwan University Hospital = 02

e.g.

| Center Nº: | 0 | 1 |
|------------|---|---|
|------------|---|---|

| Patient's | Patient's | Screening Visit |
|-----------|-----------|------------------|
| ۷°: | Initials: | Initiation Visit |

## Patients' Numbering;

Enter Patients' Group (A, B, or C), then patient's number (from 001 to 297), e.g.

|--|

## No Carbon Required (NCR) CRF

The White original and the pink NCR CRF Will be retrieved by Minapharm personnel during his / her visit to the center. The yellow NCR card will be retained by investigator folder at the site



A study population of 297 patients with compensated chronic Liver Disease, will be randomized according to fibroscan in screening visit into 2 groups:

- Group 1: with non-cirrhosis, F0, F1 and F2.
- Group 2: with advanced fibrosis and cirrhosis, F3 and F4

Subjects will be randomized into the 3 treatment groups with a balanced ratio of 1:1:1

- Group A (Experimental group), will receive Ursoplus<sup>®</sup> capsules (UDCA 250mg & Silymarin 140mg) = 99 subjects
- ➤ Group B (Control group 1), will receive Ursofalk® capsules (UDCA 250mg) = 99 subjects
- ➤ Group C (Control group 2), will receive Placebo = 99 subjects

| Patient's | Patient's | Screening Visit |
|-----------|-----------|------------------|
| Nº: | Initials: | Initiation Visit |

## **Child-Pugh Score Calculation:**

The score employs five clinical measures of liver disease. Each measure is scored 1-3, with 3 indicating most severe derangement.

| Measure | 1 point | 2 points | 3 points |
|---|---|---|---|
| Total bilirubin, µmol/l (mg/dl) | <34 (<2) | 34-50 (2-3) | >50 (>3) |
| Serum albumin, g/dl | >3.5 | 2.8-3.5 | <2.8 |
| Prothrombin time prolongation (secs) | <4.0 | 4.0-6.0 | > 6.0 |
| Ascites | None | Mild | Moderate to Severe |
| Hepatic encephalopathy | None | Grade I-II (or suppressed with medication) | Grade III-IV (or refractory) |

In primary sclerosing cholangitis (PSC) and primary biliary cirrhosis (PBC), the bilirubin references are changed to reflect the fact that these diseases feature high conjugated bilirubin levels. The upper limit for 1 point is 68  $\mu$ mol/l (4 mg/dl) and the upper limit for 2 points is 170  $\mu$ mol/l (10 mg/dl).

Chronic liver disease is classified into Child-Pugh class A to C, employing the added score from above.



| Pati<br>Nº: | ent's Patient's Initials: | Screeni<br>Initiatio | ng Visit<br>on Visit |
|---|---|---|---|
| | Screening Visit | | |
| Date | of Screening:// (DD / MMM / YYYY) | | |
| Info | med Consent: | | |
| | patient signed en consent form:// (DD / M | MM / YYYY | ) |
| | Inclusion/ Exclusion Criteria | | |
| | Inclusion Criteria | | |
| | following criteria MUST be answered YES for participant to be ided in the trial: | Yes | No |
| 1. | Male or female patient aged $\geq 18$ | | |
| 2. | Subjects with Compensated Chronic Liver Disease, defined as child 5-7. | | |
| 3. | Patients with mild disturbance of liver biochemical profile (Elevated Total Serum Bilirubin $\leq 3$ mg/dl, or elevated Direct Serum Bilirubin $\leq 2$ mg/dl, or elevated one or more of liver enzymes up to 3 times of the normal level (Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) & Gamma Glutamyl Transpeptidase (GGT)). | | |
| 4. | Non-diabetic subjects and subjects with Co<br>ntrolled DM-type 1 and 2 patients, HbA1C up to 7.5% | | |
| 5. | Non-pregnant or lactating female patients | | |
| 6. | Subjects who are willing to sign Informed Consent Form and ready to comply with the protocol for the duration of the study | | |
| | Exclusion Criteria | | |
| | following criteria MUST be answered NO for participant to be uded in the trial: | Yes | No |
| 1. | Subjects with a history of hypersensitivity to any of the ingredients of the medication being studied | | |
| 2. | Subjects with positive PCR in the past 6 months | | |
| 3. | Subjects with positive Hepatitis B surface antigen (HBsAg) | П | |

| Patie<br>Nº: | Patient's Patient's Screening Visit Initials: Screening Visit | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 4. | Subjects with elevated liver enzymes more than 3 times of the normal level (Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP) & Gamma Glutamyl Transpeptidase (GGT)). | | | | | | | | | | | |
| 5 | Subjects with Primary Biliary Cirrhosis (PBC) and Primary Sclerosing Cholangitis (PSC) | | | | | | | | | | | |
| 6 | Subjects | with | Chil | d Pug | sh Sc | ore more th | ian 7 | | | | | |
| 7 | Subjects | with | histo | ry of | blee | ding varice | S | | | | | |
| 8. | Subjects | havir | ng un | conti | ollec | l Diabetes ( | HbA1c at | ove 7 | 7.5 %) | | | |
| 9. | Subjects with any medical condition require the usage of medication may interfere with the absorption, distribution, metabolism or excretion of the drugs such as: 1- Bile acid sequestering agents such as cholestyramine and colestipol, 2- Antacids containing aluminum hydroxide. 3- Drugs affecting lipid metabolism such as estrogens, oral and hormonal contraceptives, and clofibrate (and perhaps other lipid-lowering drugs) | | | | | | | | | | | |
| 10. | | | | | | other liver<br>before stud | | | includ | ing | | |
| 11 | Subjects immune | | | | une l | iver disease | e taking c | ortico | steroic | l or | | |
| 12. | Pregnant | t or bi | east- | feedi | ng w | omen | | | | | | |
| 13 | Use of or | ral co | ntrac | eptiv | es in | child beari | ng ladies | | | | | |
| | | | | Den | ıoaı | raphic D | ata & V | ital S | Sians | <br>S | | |
| | | | | | | | | | - J | | | |
| Patie | ent Demo | grap | hy & | Vita | l Sig | ns: | | | | | | |
| Gen | der: i | Male | | | F | emale 🗌 | | | | | | |
| Birth | ndate: | / | | ' | ′ | | (DD / MM | IM / Y | YYY) | | | |
| Weig | ght: | | k | (g | | | | He | ight: | | c | :m |
| Bloo | od Pressu | ıre (S | ysto | lic/D | iasto | olic): | / | ' | | _ mm | ıHg | |

| Patient's<br>Nº: | | | Patient's<br>Initials: | | | | Screening Visit Initiation Visit |
|---|---|---|---|---|---|---|---|
| | | | Habit | S | | | |
| Smoking Hab | its: | | | | | | |
| Does the subject smoke or use tobacco products? | | | | | | | |
| How many cigarettes per day? | | | | | | | |
| Others, speci | fy: | | | | | | |
| Alcohol Consumption: | | | | | | | |
| Does the subject consume alcohol? | | | | | | | |
| If yes, how m | any units | per week? | • | | | | |
| Physical Examination | | | | | | | |
| *Please fill the noticed | relevant fo | orms of adv | erse events in | case a | ny abnoi | rmal or u | ntoward event is |
| Physical Examination | | Normal | | | Abne | ormal | |
| Findings | | | | | | | |
| Medical History | | | | | | | |
| Has the patient had any relevant medical history? | | | | | | | |

| Patient's<br>Nº: | | | | tient's<br>tials: | | | | | Screeni<br>Initiatio | |
|---|---|---|---|---|---|---|---|---|---|---|
| Condition | / illne | ess /surgic | al procedure | е | | | | | o date<br>MM/YYYY) | Or tick if ongoing ? |
| | | | | | | / | - - | / | | |
| | | | | | | | - | / | | |
| | | | | | | / | _ | I | | |
| Is the participant taking any concomitant medications? If Yes: Complete Concomitant Medication Page 26 Abdominal Ultrasound | | | | | | | | | | |
| Date of Ultrasound:/ (DD / MMM / YYYY) | | | | | | | | | | |
| Liver | | Normal Abnormal | | | | | | | | |
| lf abnormal,<br>findings: | , | Portal Vein Diameter:mm (N. up to 14mm) | | | | | | | | |
| | | Ascites: | ☐ No | Y | 'es | If yes, | Amoι | ınt: | | |
| Spleen | | Normal | | | Abnormal | | | | | |
| lf abnormal,<br>findings: | , | | | | | | | | | |
| illidiligs. | | Splenic V | ein Diamete | er: | ••••• | mm | | | | |
| Gall Bladder | r | Normal | | | | Abno | rmal | | | |
| lf abnormal,<br>findings: | , | Common | Bile Duct (C | BD) Dia | meter: | | | (N. u | p to 6mm | ) |

| Patient's<br>Nº: | | Patient'<br>Initials: | s | | | Screening Visit<br>Initiation Visit |
|---|---|---|---|---|---|---|
| Vibration-cor | ntrolled tra | nsient ela | sto | graphy | with C | AP (Fibroscan) |
| Date of Fibroscan: | Date of Fibroscan:/ (DD / MMM / YYYY) | | | | | |
| | Liver stiffne | ss measurem | ent | | Fibroscan score | |
| Liver | | ☐ F0/I | | | | /F1 |
| If abnormal,<br>findings: | | | | | | |
| | Sat | fety Laboi | rato | ry Tes | ts | |
| Date of Laboratory Tests:// (DD / MMM / YYYY) | | | | | | |
| Laboratory Param | neter | Value | Unit | | If parameter indicated as out of normal range on report, please check if clinically significant: | |
| ALT | | | | | ☐ No | ☐ Yes |
| AST | | | | | □ No | ☐ Yes |
| Alkaline Phospha | tase (ALP) | | | | ☐ No | ☐ Yes |
| Gamma-GT | | | | | ☐ No | ☐ Yes |
| Total Bilirubin | | | | | ☐ No | ☐ Yes |
| Direct bilirubin | | | | | ☐ No | ☐ Yes |
| S Albumin | | | | | ☐ No | ☐ Yes |
| PT | | | | | ☐ No | ☐ Yes |
| HbA1c for diabeti | c patients | | | | ☐ No | ☐ Yes |
| PCR/ Antibody for | r hepatitis C | | | | ☐ No | ☐ Yes |
| HBs Ag | | | | | □No | ☐ Yes |
| Serum β-HCG (for child bearing peri | | | | | ☐ No | ☐ Yes |

| Patie<br>Nº: | Patient's Patient's Screening Visit Initials: Screening Visit Initiation Visit | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Assess | men | t for o | quality | of life ( | The RA | ND 36 | 6-Iten | n Hea | lth S | urvey | ) |
| | Comple | eted | | | | No | ot Com | pleted | 1 | | | |
| | | | | En | d of So | roonin | a Vioi | | | | | |
| | | | | EIII | <i>a</i> 01 30 | reenin | y visi | | | | | |
| End | End of Screening Visit Checklist: Yes No | | | | | | | | | | | |
| Does the participant meet the inclusion and exclusion criteria to date? | | | | | | to | | | | | | |
| 2. | 2. Have all Screening Visit procedures been completed? | | | | | | | | | | | |
| 3. | 3. Have the Medical History and Concomitant Medication pages been completed? | | | | | | | | | | | |
| Parti | cipant's e | ligibil | ity: | | | | | | | | | |
| Is the | participan | nt eligil | ole to ta | ake part ir | the Clini | cal Study? | | | | | | |
| ☐ Ye | es | | | | | | | | | | | |
| □ No | o, Please g | give re | ason fo | or screen | failure bel | ow | | | | | | |
| Reas | on(s) for | screei | n failur | e: | | | | | | | | |
| 1. | | | | | | | | | | | | |
| 2. | | | | | | | | | | | | |
| Inves | stigator Si | gn-Of | f | | | | | | | | | |
| | stigator's l | | | | | <br>Date : | | / _<br>// MM / Y | | _ | | |

| Patient's<br>Nº: | | Patient's<br>Initials: | | | eening Visit<br>tiation Visit |
|---|---|---|---|---|---|
| | | Randomiz | ation | | |
| Group A | | Group B | | Group C | |
| Drug Dispense | | | | | |
| Date of Drug Dispense:// (DD / MMM / YYYY) | | | | | |
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | | | | |
| | | | | 1 | |
| Drug D | ispense | Number | of Capsules | Number | Number of Blisters |
| Drug A | , B, or C | | | | |
| Investigator's Name: | | | | | |
| Investigator's Sign | ature: | Dat | e:/ | | |
| | | | (DD/MMM/ | 1111) | |

| Patient's<br>N°: | | Patient's<br>nitials: | | Visit 2 (Week 4)<br>Follow Up Visit<br>1 |
|---|---|---|---|---|
| Visit 2 (Week 4) (may be done by phone call) | | | | |
| Date of Visit 2:// (DD / MMM / YYYY) | | | | |
| | , | Vital Signs | | |
| Vital Signs & Weight: | | | | |
| Weight: | Kg | | | |
| Blood Pressure (Systolic/Diastolic):/ mmHg | | | | |
| Physical Examination | | | | |
| *Please fill the relevant forms of adverse events in case any untoward or unusual event that occurred since last visit, whether it is believed to be related to the study drug or not. | | | | |
| Physical<br>Examination | Normal | | Abnormal | |
| Findings | | | | |
| | Dr | ug Dispense | | |
| Date of Drug Dispense:// (DD / MMM / YYYY) | | | | |
| Drug | g Dispense | Number of Caps | ules Num | ber of Blisters |
| Druç | g A, B, or C | | | |

| Patient's<br>Nº: | | atient's<br>itials: | Visit 2 (Week 4) Follow Up Visit 1 |
|---|---|---|---|
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | | |
| Is the participant taking any concomitant medications? No | | | |
| Is the participant had any Adverse Events The investigator shall ask probing questions, allowing | | | |
| the patient that occurre patient) beli | The investigator shall ask probing questions, allowing the patient to tell about any untoward or unusual event that occurred since the last visit, whether he/she (the patient) believes it is related to the study drug or not? (including abnormal physical examination/ laboratory results) | | |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | | |
| Investigator's Name: | | | |
| Investigator's S | ignature: | Date: / / | |
| | | (DD / MMM / YYYY) | |

| Patient's<br>Nº: | | Patient's<br>Initials: | | visit 3 (Week 8) ollow Up Visit 2 |
|---|---|---|---|---|
| Visit 3 (Week 8) (may be done by phone call) | | | | |
| Date of Visit 3:// (DD / MMM / YYYY) | | | | |
| | | Vital Signs | | |
| Vital Signs & Weight: | | | | |
| Weight: | <b>Weight</b> : Kg | | | |
| Blood Pressure (Systolic/Diastolic):/mmHg | | | | |
| Physical Examination | | | | |
| *Please fill the relevant forms of adverse events in case any untoward or unusual event that occurred since last visit, whether it is believed to be related to the study drug or not. | | | | |
| Physical<br>Examination | Normal | | Abnormal | |
| Findings | Examination | | | |
| | Drug Dispense | | | |
| Date of Drug Dispense:/ (DD / MMM / YYYY) | | | | |
| Drug | Dispense | Number of Caps | ules Numb | per of Blisters |
| Drug | A, B, or C | | | |

| Patient's<br>Nº: | | Patient's Initials: | Visit 3 (Week 8)<br>Follow Up Visit 2 |
|---|---|---|---|
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | | |
| Is the participant taking any concomitant medications? No | | | |
| Is the participant had any Adverse Events | | | |
| The investigator shall ask probing questions, allowing the patient to tell about any untoward or unusual event that occurred since the last visit, whether he/she (the patient) believes it is related to the study drug or not? (including abnormal physical examination/ laboratory results) | | | |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | | |
| Investigator's N | ame: | | |
| Investigator's S | ignature: | Date://///// | |

| Patient's<br>Nº: | | Patient'<br>s<br>Initials: | | Visit 4 (Week 12)<br>Follow Up Visit 3 |
|---|---|---|---|---|
| | Visit 4 (Week 12) | | | |
| Date of Visit 4: | Date of Visit 4:// (DD / MMM / YYYY) | | | |
| | | Vital Sig | ns | |
| Vital Signs & | Weight: | | | |
| Weight: | Kg | | | |
| Blood Pressu | Blood Pressure (Systolic/Diastolic):/mmHg | | | |
| | Phy | sical Exar | nination | |
| *Please fill the relevant forms of adverse events in case any untoward or unusual event that occurred since last visit, whether it is believed to be related to the study drug or not. | | | | |
| Physical<br>Examination | Normal | | Abnormal | |
| Findings | | | | |
| | Assess | ment for q | uality of life | |
| The RAND 36-Item Health Survey | | | | |
| Comple | | | Not Completed | |

| Patient's<br>Nº: | | Patient'<br>s<br>Initials: | | | | Visit 4 (W<br>Follow U | , |
|---|---|---|---|---|---|---|---|
| | Di | rug Disp | ense | | | | |
| Date of Drug Dispe | ense:/ | _/ | _ (DD/N | имм / \ | YYYY) | ) | |
| Drug Di | spense | Number | of Capsu | les | Nu | mber of B | listers |
| Drug A, | B, or C | | | | | | |
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | | | | | | |
| Is the participant taking any concomitant medications? Is the participant taking any Page 26 | | | | | dication | | |
| ls the participant | had any Advers | e Events | | | | | |
| The investigator the patient to tel that occurred sin patient) believes (including abnormsults) | Il about any unto<br>nce the last visit<br>s it is related to t | ward or u<br>, whether<br>he study | inusual (<br>he/she (<br>drug or i | event<br>the<br>not? | | ☐ <b>No</b><br><b>If Yes:</b> Co<br>Page | • |
| I have updated the severity and outcom study information ob | ne and confirm that | , to the bes | | | | | |
| Investigator's Name: | · | | | | | | |
| Investigator's Signat | ture: | Date | :/ | /_ | | _ | |
| | | | (DD / M | MM / YY | YY) | | |

| Patient's<br>Nº: | | Patient'<br>s<br>Initials: | | Visit 5 (Week 16)<br>Follow Up Visit 4 |
|---|---|---|---|---|
| , | Visit 5 (Week 16) | (may be done by | phone | call) |
| Date of Visit 5:// (DD / MMM / YYYY) | | | | |
| | , | Vital Signs | | |
| Vital Signs & Weight: | | | | |
| Weight: | Kg | | | |
| Blood Pressure (Systolic/Diastolic):/mmHg | | | | |
| Physical Examination | | | | |
| | *Please fill the relevant forms of adverse events in case any untoward or unusual event that occurred since last visit, whether it is believed to be related to the study drug or not. | | | |
| Examination | Normal | | Abnormal | |
| Findings | | | | |
| | | Dianana | | |
| | Dr | ug Dispense | | |
| Date of Drug D | ispense:/ | _/ (DD / MM | MM / YYYY) | |
| Dru | g Dispense | Number of Capsule | es Nur | nber of Blisters |
| Dru | ıg A, B, or C | | | |

| Patient's | Patient' s nitials: | Visit 5 (Week 16)<br>Follow Up Visit 4 |
|---|---|---|
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | |
| Is the participant taking any concomitant medications? | ☐ <b>No If Yes:</b> Complete Con Page | |
| Is the participant had any Adverse Events The investigator shall ask probing questions, allowing | | |
| the patient to tell about any untow<br>that occurred since the last visit,<br>patient) believes it is related to th<br>(including abnormal physical exa<br>results) | ward or unusual event<br>whether he/she (the<br>e study drug or not? | ☐ No ☐ Yes If Yes: Complete Page 30 |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | |
| Investigator's Name: | | |
| Investigator's Signature: | Date: / | |

| Patient's<br>Nº: | | Patient' | | Visit 6 (Week 20)<br>Follow Up Visit 5 |
|---|---|---|---|---|
| L | | iriiliais. [ | | |
| Visit 6 (Week 20) (may be done by phone call) | | | | |
| Date of Visit 6:// (DD / MMM / YYYY) | | | | |
| Vital Signs | | | | |
| Vital Signs & Weight: | | | | |
| Weight: | Kg | | | |
| Blood Pressu | re (Systolic/Diastolic) | :/ | mn | nHg |
| | Phys | ical Examinatio | n | |
| occurred since la | elevant forms of advers | | | |
| Examination | | _ | | _ |
| Findings | | | | |
| | Dı | rug Dispense | | |
| Date of Drug Di | spense:/ | _/ (DD/N | MMM / YYYY) | |
| Drug | g Dispense | Number of Capsu | iles Nun | ber of Blisters |
| Dru | g A, B, or C | | | |

| Patient's<br>Nº: | | ient'<br>s<br>ials: | Visit 6 (Week 20)<br>Follow Up Visit 5 |
|---|---|---|---|
| Drugs are dispensed for the patient to be sufficient for 30 days of treatment The subject is asked to take the treatment daily and come next visit with the empty blisters after 30 days, with a window of 7 days. | | | |
| - | ipant taking any<br>t medications? | ☐ <b>No If Yes:</b> Complete Cor | |
| Is the participant had any Adverse Events | | | |
| the patient that occurre patient) beli | gator shall ask probing of<br>to tell about any untowal<br>ed since the last visit, where<br>eves it is related to the<br>bnormal physical exam | rd or unusual event<br>hether he/she (the<br>study drug or not? | ☐ No ☐ Yes If Yes: Complete Page 30 |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | | |
| Investigator's N | lame: | | |
| Investigator's S | signature: | Date:/// [DD / MMM / YYYY] | - <b></b> |

| Patient's N°: | Patie<br>Initia | | En | d of Study Visit<br>(Week 24) |
|---|---|---|---|---|
| End of study Date of End of study visit:/ (DD / MMM / YYYY) | | | | |
| Vital Signs | | | | |
| Vital Signs & Weight: | Vital Signs & Weight: | | | |
| <b>Weight</b> : Kg | | | | |
| Blood Pressure (Systolic/ | Diastolic): | / | mmHg | |
| | Physical Examination | | | |
| *Please fill the relevant forms since last visit, whether it is b | | - | | t that occurred |
| Physical Examination | Normal | | Abnormal | |
| Findings | | | | |
| G | | | | |
| | Assessment t | or quality of | life | |
| | | or quality of l | | |

| Patient's N°: | | ent's<br>als: | | End of Study Visit<br>(Week 24) |
|---|---|---|---|---|
| Safety Laboratory Tests | | | | |
| Date of Laboratory Tests:// (DD / MMM / YYYY) | | | | |
| Laboratory Parameter | Value | Unit | If parameter indicated as out of normal range on report, please check if clinically significant: | |
| ALT | | | □ No | ☐ Yes |
| AST | | | ☐ No | ☐ Yes |
| Alkaline Phosphatse (AL | P) | | ☐ No | ☐ Yes |
| Gamma-GT | | | ☐ No | Yes |
| S.Albumin | | | □No | Yes |
| Total Bilirubin | | | ☐ No | Yes |
| Direct bilirubin | | | ☐ No | Yes |
| Serum β-HCG (for Female with child bearing potent only) | | | □No | ☐ Yes |
| | | · | · | |
| Vibration-cont | rolled transient | elastograp | hy with CA | P (Fibroscan) |
| Date of Fibroscan:/_ | /( | DD / MMM / YYYY) | ) | |
| | Liver stiffness me | asurement | Fibr | oscan score |
| Liver | | ☐ F0/F1 ☐ F2 ☐ F3 ☐ F4 | | |
| If abnormal, findings: | | | | |
| Is the participant taking any Oncomitant medications? | | | | |

| Patient's Nº: | | Patient's<br>Initials: | | Study Visit<br>ek 24) |
|---|---|---|---|---|
| If Yes: Complete Concomitant Medication Page 26 | | | | |
| Is the participant had any Adverse Events | | | | |
| The investigator shall ask probing questions, allowing the patient to tell about any untoward or unusual event that occurred since the last visit, whether he/she (the patient) believes it is related to the study drug or not? (including abnormal physical examination/ laboratory results) | | | | |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | | | |
| Investigator's Nam | ne: | | | |
| Investigator's Sigr | nature: | | _ / /<br>DD / MMM / YYYY | |

| Patient's Nº: | | | | | Pati | ent's Initials: | |
|---|---|---|---|---|---|---|---|
| Concomitant Medication Form | | | | | | | |
| Medication (Record Generic or trade name) | Reason for use<br>(Medical History<br>diagnosis or other<br>reason, e.g.<br>Prophylaxis) | Dose<br>and<br>units | Frequency | Route | Start Date<br>(DD/MMM/YYYY) | Stop Date (DD//MMM/YYY) | Or tick<br>if<br>ongoing |
| 1. | | | | | | | |
| 2. | | | | | | | |
| 3. | | | | | | | |
| 4. | | | | | | | |
| 5. | | | | | | | |
| 6. | | | | | | | |
| 7. | | | | | | | |
| PI signature | | | | Date: _ | | | |

| Pat | tient's Nº: | | | | | | | Pa | tient's Initials: | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Adverse Events (1/2) | | | | | | | | | | | |
| | | | | | | | 1 | T | | | | |
| AE<br>No | <b>Event Name</b><br>(Please give Diagno<br>known) | Start da<br>(DD/MMM/\ | | Stop date<br>(DD/MMM/YYYY) | Serious? | Con-<br>comitant<br>Medication<br>given | Severity<br>0 - Mild<br>1- Mode-<br>rate<br>2 - Severe | Study Drug Action 0 - None 1 - Temporarily Interrupted 2 - permanently withdrawn | Outcome 1- Death related to AE 2- Not resolved/Not recovered 3- Resolved/ Recovered 4- Resolved/ Recovered with Sequelae 5- Resolving/ Recovering 6- Unknown | Relation<br>Study D<br>0 - Certain<br>1 – Probab<br>2 - Possible<br>3 - Unlikely<br>4 – Conditi<br>Unclassifie<br>5 - Un-asse<br>Unclassifia | rug lle/Likely e onal/ d essable/ | • |
| | | | | | ☐ No | ☐ No | | | | | | |
| 1 | | /_ | <u></u> | | ☐ Yes | Yes | | | | | | |
| 2 | | I | _I | | ☐ No<br>☐ Yes | ☐ No<br>☐ Yes | | | | | | |
| 3 | | / | _I | | ☐ No | ☐ No<br>☐ Yes | | | | | | |
| 4 | | | <u></u> | | ☐ No | ☐ No | | | | | | |
| 5 | | | | | ☐ No | ☐ No<br>☐ Yes | | | | | | |
| | | | | d have assessed t<br>ly information obta | | | sality, sev | erity and οι | itcome and confirm t | hat, to the | e best of | f my |
| | PI signature _ | | | | | Date: | | | | | | |

| Pat | tient's Nº: | | | | | | Pat | tient's Initials: | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Ad | verse Ev | /ents (2/2 | 2) | | | |
| AE<br>No | <b>Event Name</b><br>(Please give Diagnosis if<br>known) | Start date<br>(DD/MMM/YYYY) | Stop date<br>(DD/MMM/YYYY) | Serious? | Con-<br>comitant<br>Medication<br>given | Severity<br>0 - Mild<br>1- Mode-<br>rate<br>2 - Severe | Study<br>Drug<br>Action<br>0 - None<br>1 -<br>Temporarily<br>Interrupted<br>2 -<br>permanently<br>withdrawn | Outcome 1- Death related to AE 2- Not resolved/Not recovered 3- Resolved/ Recovered 4- Resolved/ Recovered with Sequelae 5- Resolving/ Recovering 6- Unknown | Relationship to<br>Study Drug<br>0 - Certain<br>1 - Probable/Likely<br>2 - Possible<br>3 - Unlikely<br>4 - Conditional/<br>Unclassified<br>5 - Un-assessable/<br>Unclassifiable |
| 4 | | | | ☐ No | ☐ No | | | | |
| 1 | | | / | Yes | Yes | | | | |
| 2 | | | | ☐ No<br>☐ Yes | ☐ No<br>☐ Yes | | | | |
| 3 | | | | ☐ No | ☐ No | | | | |
| 4 | | | | ☐ No | ☐ No<br>☐ Yes | | | | |
| 5 | | | | ☐ No | ☐ No | | | | |
| | I have reviewed the knowledge, it accura | | | | | usality, sev | erity and ou | tcome and confirm | that, to the best of my |
| | PI signature | | | | Date: _ | | | | |

| Patient's<br>Nº: | | | | | Patie<br>Initi | ent's<br>als: | | | | | Un | sched | uled Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Unscheduled Visit | | | | | | | | | | | | | | |
| Date of Unsch | edul | ed Vi | isit: | / | ' — — — | _/ | | . (DI | D / MM | 1M / Y | YYY | ) | | _ |
| | | | | | Vit | al Si | gns | | | | | | | |
| Vital Signs & | Wei | ght: | | | | | | | | | | | | |
| Weight: | | l | <b>K</b> g | | | | | | | | | | | |
| Blood Pressure (Systolic/Diastolic):/ mmHg | | | | | | | | | | | | | | |
| | | | | Ph | ysica | I Ex | amin | atio | n | | | | | |
| *Please fill the occurred since | | | | | | | | _ | | | | | | _ |
| Physical<br>Examination | | | Norm | | | | | | Abno | | | | | |
| Findings | | | | | | | | | | | | | | |
| Is the partic | • | | _ | - | | ☐ No ☐ Yes If Yes: Complete Concomitant Medication Page 26 | | | | _ | | | | |
| Is the particip | oant | had | any | Adv | erse E | vents | \$ | | | | | | | _ |
| The investigator shall ask probing questions, allowing the patient to tell about any untoward or unusual event that occurred since the last visit, whether he/she (the patient) believes it is related to the study drug or not? (including abnormal physical examination/ laboratory | | | | | | | | | | | | | | |
| I have updated the AEs on page And have assessed them for seriousness, causality, severity and outcome and confirm that, to the best of my knowledge, it accurately reflects the study information obtained for this participant: | | | | | | | | | | | | | | |
| Investigator's N | ame: | _ | | | | _ | | | | | | | | |
| nvestigator's Signature: Date:/(DD / MMM / YYYY) | | | | | | | | | | | | | | |

| Patient's<br>Nº: | Patient's Initials: | Study Completion page |
|---|---|---|
| Study Completion | | |

| Did participant complete the trial? | |
|---|---|
| Yes, Please provide date of last day: | |
| //20(DD/ | MMM / YYYY) |
| No, Please provide date of withdrawal and complete belo | w: |
| //20(DD/ | MMM / YYYY) |
| Early Withdrawal: please tick most appropriate reason for participant not completing the trial: | |
| Adverse Events related: please state related AE: _ | (add details to |
| AE page) | |
| ☐ Participant's decision, specify: | |
| ☐ Investigator's decision, specify: | |
| ☐ Sponsor's decision | |
| ☐ Lost to follow up | |
| ☐ Patient deceased | |
| $\square$ Ineligibility (either arising during the study o screening) | r retrospective having been overlooked at |
| ☐ Significant protocol deviation | |
| ☐ Significant non-compliance with treatment re | egimen or study requirements |
| ☐ Disease progression which requires discont inability to continue to comply with study process. | inuation of the study medication or results in edures |
| Consent withdrawn. | |
| ☐ Pregnancy or discontinuation of contracepti | on |
| Other, specify: | _ |
| Investigator Sign off | |
| Investigator's Name: | |
| Investigator's Signature: | Date :// (DD / MMM / YYYY) |